CLINICAL TRIAL: NCT01472666
Title: Dairy Lipids, Proteins, and the Metabolic Syndrome - "DairyHealth"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Arla Foods (Industry); Wageningen University (Other); University of Dublin, Trinity College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CERN-DairyHealth
Record Dates: First submitted 2011-11-01; First posted 2011-11-16 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2013-07

CONDITIONS: Metabolic Syndrome; Type 2 Diabetes; Cardiovascular Disease; Abdominal Obesity
Keywords: Medium chain fatty acids; Saturated fatty acids; Whey protein; Casein protein; Metabolic syndrome; Type 2 diabetes; Cardiovascular disease; Dairy products; Dietary intervention
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Obesity, Abdominal | interventions — Whey; Caseins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fat rich in MC-SFA (Experimental): 63 gram milk fat with high content of MC-SFA (C6-C12=8.5 g) incorporated in rolls, muffin and as butter.
  Interventions: Dietary Supplement: High content of MC-SFA
- Fat low on MC-SFA (Experimental): 63 gram milkfat with low content of MC-SFA (C6-C12=6.9 g) incorporated in rolls, muffin and as butter
  Interventions: Dietary Supplement: Low content of MC-SFA
- Casein protein (Experimental): 60 gram casein protein (Miprodan 30) ingested twice daily with 600 ml water.
  Interventions: Dietary Supplement: Casein
- Whey protein (Experimental): 60 gram whey protein (Lacprodan DI-9224) ingested twice daily with 600 ml water.
  Interventions: Dietary Supplement: Whey

INTERVENTIONS:
Dietary Supplement: High content of MC-SFA — 12 weeks dietary intervention
  Arms: Fat rich in MC-SFA
Dietary Supplement: Whey — 12 weeks dietary intervention
  Arms: Whey protein
Dietary Supplement: Low content of MC-SFA — 12 weeks dietary intervention
  Arms: Fat low on MC-SFA
Dietary Supplement: Casein — 12 weeks dietary intervention
  Arms: Casein protein

SUMMARY:
Dairy food contains a large amount of long-chain saturated fat, which traditionally has been linked to increased risk of cardiovascular disease (CVD). However, recent data indicates a more neutral role. Milk fat contains large amounts of medium-chain saturated fatty acids (MC-SFA), which may have beneficial effects on human health. In addition, milk proteins and in particular whey proteins have been shown to have a beneficial effect on glucose disposal as well as anti-inflammatory properties. Therefore dairy products have a potential role in the treatment of the metabolic abnormalities of metabolic syndrome (MeS). However, human data from intervention studies are lacking.

Aims of this project is to explore and understand the influence on human health of both medium-chain saturated fatty acids from milk fat and bioactive milk proteins per se as well as their interaction and potential positive synergy on the MeS.

The investigators hypothesize that whey protein and medium-chain saturated fatty acids improve insulin sensitivity, postprandial lipid metabolism, blood pressure and inflammatory stress in humans and that they possess preventive effects on the risk of developing CVD and type 2 diabetes mellitus (T2DM).

A total of 64 people with MeS or abdominal obesity will be included. The design is a randomized double-blinded, controlled parallel diet-intervention trial.

Subjects are assigned one of four experimental diets for 12 weeks. The diets consist of either a diet with low levels of MC-SFA + whey protein (LF + whey), a diet high in MC-SFA + whey protein (HF + whey), a diet high in MC-SFA + casein protein (HF + casein) or a diets with low levels of MC-SFA + casein protein (LF + casein). The subjects are advised how to integrate the test foods in their habitual diet, which also continues unchanged. The subjects' energy intake is matched so they are kept weight stable throughout the study.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

Metabolic syndrome

* Central obesity (Waist: female ≥ 80 cm; male ≥ 94 cm)
* with two or more of the following
* Fasting triglyceride > 1.7 mmol/l
* HDL-cholesterol; male < 1.03 mmol/l, female < 1.29 mmol/l
* BP ≥ 130/85
* Fasting plasma glucose ≥ 5,6 mmol/l (but not diabetes)

Or abdominal obesity (Waist: female ≥ 80 cm; male ≥ 94 cm)

Exclusion Criteria:

* Significant cardiovascular, renal or endocrine disease
* Psychiatric history
* Treatment with steroids
* Alcohol- or drug-addiction
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Postprandial triglyceride response | Change from week 0 to week 12
  Compare the changes in mean difference of 6 hours incremental area under the curve (iAUC) (week 12 - week 0) between the groups and the intervention components.

SECONDARY OUTCOMES:
24 hour blood pressure (BP) | Change from week 0 to week 12
  Spacelabs, model 90207/90217, USA
Indirect calorimetry | Change from week 0 to week 12
  Measured 2 times during meal test.
Dexa-scan (body composition) | Change from week 0 to week 12
  Total body fat percentage, lean mass, gynoid, and android fat percentage, and total body weight.
Weight | Change from week 0 to week 12
Biomarkers in blood samples | Change from week 0 to week 12
  Glucose, insulin, glucagon, HbA1c. free fatty acids, Lipid profile (total-cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglyceride). Inflammations markers (interleukin-6 (IL-6), interleukin-10 (IL-10), interleukin-1 receptor antagonist (IL-1RA), interleukin-1 beta (IL-1b), high sensitive c-reactive protein (hs-CRP), adiponectin, monocyte chemoattractant protein-1 (MCP-1), Rantes (CCL5)). Incretins (GLP-1, GIP). Nutrigenomics. Metabolomics. Proteomics.
Waist and hip circumference | Change from week 0 to week 12
Fat tissue biopsy | Change from week 0 to week 12
  Fat tissue gene expression. Twice during meal test.
Biomarkers in urine | Change from week 0 to week 12
  Nutrigenomics and metabolomics
Glucose tolerance | Change from week 0 to week 12
  Oral glucose tolerance test (OGTT) (with insulin and glucose measurement at time -15 min, -10 min, 0 min, 30 min, 60 min, and 120 min). Hereby calculating the homeostatic model assessment of insulin resistance (HOMA-IR) and the Matsuda index.
Dietary compliance | Change from week 0 to week 12
  3-day food diary.
Postprandial apolipoprotein-48 (apoB-48), 6 hour | Change from week 0 to week 12
  Meal test, blood samples at time 0,2,4 and 6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Hermansen, Professor, Principal Investigator — Aarhus University Hospital; Hanne C Bertram, Scientist, Study Chair — Department of Food Science, University of Aarhus; Lorraine O'Driscoll, Professor, Study Chair — School of Pharmacy & Pharmaceutical Sciences, Trinity College Dublin, Ireland; Michael Müller, Professor, Study Chair — Division of Human Nutrition, Wageningen University, The Netherlands
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Derived] Bohl M, Bjornshave A, Rasmussen KV, Schioldan AG, Amer B, Larsen MK, Dalsgaard TK, Holst JJ, Herrmann A, O'Neill S, O'Driscoll L, Afman L, Jensen E, Christensen MM, Gregersen S, Hermansen K. Dairy proteins, dairy lipids, and postprandial lipemia in persons with abdominal obesity (DairyHealth): a 12-wk, randomized, parallel-controlled, double-blinded, diet intervention study. Am J Clin Nutr. 2015 Apr;101(4):870-8. doi: 10.3945/ajcn.114.097923. Epub 2015 Jan 14. PMID 25833983